CLINICAL TRIAL: NCT03577821
Title: Surgical Modalities and Early Outcome of Total Arterial Revascularization in CABG
Brief Title: Early Outcome of Total Arterial Revasclarization in IHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hosam mohamed farouk, Assistant lecturer cardiac surgery, Assiut University
Other Study IDs: arterial revascularization
Record Dates: First submitted 2018-06-08; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complete arterial coronary artery bypass grafting (CABG) is a surgical option to improve long-term results in the treatment of coronary artery disease (CAD). The goal of coronary artery bypass operations is complete revascularization and there is an increasing interest toward complete arterial revascularization to achieve this goal because of high late failure of saphenous vein graft

DETAILED DESCRIPTION:
The availability of arterial conduit which is long enough to perform complete arterial revascularization is the limitation of the procedure and it is mandatory to adjust length of the available graft to serve the need. To overcome this problem, sequential or/ and composite grafting techniques are used and one conduit is used for more than one distal anastomoses or multiple arterial grafts are preferred. Bilateral internal mammarian arteries (IMAs), the gastroepiploic artery (GEA), inferior epigastric artery and the radial artery (RA) have been used as conduits in selected patients. However, sequential grafting using arterial grafts may not be convenient for all circumstances and sometimes surgical technique may be challenging. Besides, classical Y-graft technique of RA has the disadvantage of shortening the graft. Harvesting multiple arterial conduits is more time consuming and may result in elevated operative trauma and perioperative complications (sternal dehiscence, sternal infection, pulmonary complications, required laparatomy, prolonged ICU time and hospitalization time, etc.). Every eligible patient should receive total arterial revascularization, the cornerstone of which is BITA grafting. Patients with a body mass index (BMI) of over 35, diabetes or severe airway disease or who are undergoing radio- therapy or immunosuppression are only relatively contra- indicated for BITA use.7 If more conduits are required, the RA can be prepared at the same time as the LITA, and its harvesting is associated with favorable early outcomes Prior to harvesting, a modified Allen test is performed. If a hyperemic response to the previous ischemic hand is noticed within 5 s, the collateral ulnar circulation is adequate. Restoration of the blood circulation to the ischemic hand later than 10 s after the ulnar release excludes the RA from being used.

Duplex examination and pulse oximetry can also be used to preoperatively evaluate the RA and ulnar artery. Moreover, the RA should be avoided when cardiac catheterization has been recently pre- ceded by injuring the vessel and when the RA might be used for future fistulae in patients who are receiving or who are likely to receive dialysis] RAs less than 2 mm in diameter are also avoided due to the possibility of vasospasm.

Finally, the extent of stenosis of the target coronary vessel may also constitute a contraindication for arterial conduit use due to competitive flow. Hence, stenoses of less than 70% in the left coronary bed and less than 90% in a dominant right coronary artery should prevent the use of an arterial graft.

ELIGIBILITY:
Inclusion Criteria:

All patients who will undergo total arterial revascularization either with single or multi vessel coronary artery disease are to be put in the investigator's study work.

-

Exclusion Criteria:

* there is no any.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who will be operated in cardiothoracic surgey department Assiut university hospital from July 2018 to december 2019 by performing total arterial revascularization (CABG) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
target vessel revascularization | baseline-3 months
  readmission for revascularization due to graft failure

SECONDARY OUTCOMES:
Major cardiac events | baseline-3 months
  (myocardial infarction, stroke, readmission for CHF)
Postoperative morbidity | 3 months
  frequency of peroperative/ postoperative complications according to registration schemes
Wound infection | 3 months
  Readmission for wound infection (superficial sternal wound infection, deep sternal wound infection, saphenous vein related wound infection, need for VAC therapy, need for surgical debridment, need for prolonged antibiotic therapy)
Bleeding | Early postoperative up to 1 week
  surgical bleeding requiring re-exploration
Length of ICU stay | Early postoperative up to 1 week
  number of days in ICU

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doshi R, Rao G, Shlofmitz E, Donnelly J, Meraj P. Comparison of In-Hospital Outcomes After Percutaneous Revascularization for Peripheral Arterial Disease in Patients With a Body Mass Index of >30 kg/m2 Versus </=30 kg/m2 (from the National Inpatient Sample). Am J Cardiol. 2017 Nov 1;120(9):1648-1652. doi: 10.1016/j.amjcard.2017.07.065. Epub 2017 Jul 31. PMID 28842147
- [Background] Raja SG, Ilsley C, De Robertis F, Lane R, Kabir T, Bahrami T, Simon A, Popov A, Dalby MC, Mason M, Grocott-Mason R, Smith RD, Iqbal MB. Mid-to-long term mortality following surgical versus percutaneous coronary revascularization stratified according to stent subtype: An analysis of 6,682 patients with multivessel disease. PLoS One. 2018 Feb 6;13(2):e0191554. doi: 10.1371/journal.pone.0191554. eCollection 2018. PMID 29408926
- [Background] Schwann TA, Tatoulis J, Puskas J, Bonnell M, Taggart D, Kurlansky P, Jacobs JP, Thourani VH, O'Brien S, Wallace A, Engoren MC, Tranbaugh RF, Habib RH. Worldwide Trends in Multi-arterial Coronary Artery Bypass Grafting Surgery 2004-2014: A Tale of 2 Continents. Semin Thorac Cardiovasc Surg. 2017 Autumn;29(3):273-280. doi: 10.1053/j.semtcvs.2017.05.018. Epub 2017 Aug 8. PMID 29195570
- [Background] Buttar SN, Yan TD, Taggart DP, Tian DH. Long-term and short-term outcomes of using bilateral internal mammary artery grafting versus left internal mammary artery grafting: a meta-analysis. Heart. 2017 Sep;103(18):1419-1426. doi: 10.1136/heartjnl-2016-310864. Epub 2017 Jun 23. PMID 28646103
- [Background] Saraiva J, Antunes PE, Antunes MJ. Coronary artery bypass surgery in young adults: excellent perioperative results and long-term survival. Interact Cardiovasc Thorac Surg. 2017 May 1;24(5):691-695. doi: 10.1093/icvts/ivw407. PMID 28453797